CLINICAL TRIAL: NCT01492972
Title: Phase III Study of Image Guided Radiation Therapy With or Without Androgen Suppression for Intermediate Risk Adenocarcinoma of the Prostate
Brief Title: Hypo-fractionated Radiation Therapy With or Without Androgen Suppression for Intermediate Risk Prostate Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Proton Collaborative Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GU003-10
Record Dates: First submitted 2011-12-09; First posted 2011-12-15 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
Keywords: Prostate; proton; radiation; intermediate risk
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiation; Leuprolide; Goserelin; Buserelin; Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radiation Alone (Active Comparator): Proton Radiation Total Dose=70 Gy(RBE) OR High Dose Radiation with IMRT Alone=81 Gy OR Intraoperative LDR Brachytherapy and IMRT=45 Gy
  Interventions: Radiation: Radiation
- Radiation + Androgen Suppression (Experimental): Androgen Suppression Therapy x 6 months + Radiation
  Interventions: Radiation: Radiation; Drug: Androgen Suppression Therapy

INTERVENTIONS:
Radiation: Radiation — Consists of:
  1. Conformal Proton Radiation Dose: 2.5 Gy (RBE) five days a week in 28 treatments over 5.5-6.5 weeks (total dose: 70 Gy (RBE))
  2. High Dose Radiation with IMRT alone: 1.8 Gy five days a week in 45 treatments over 9-10 weeks (total dose: 81 Gy)
  3. Intraoperative LDR Brachytherapy and IMRT: 100Gy Pad103 implant and IMRT 1.8 Gy five days a week in 25 treatments over 5-6 weeks (total dose: 45 Gy)
Drug: Androgen Suppression Therapy — Androgen suppression will begin 8 - 10 weeks prior to the start of RT for a total of 6 (+/- 2) months. Luteinizing Hormone-Releasing Hormone (LHRH) agonist therapy will consist of analogs approved by the FDA (or by Health Canada for Canadian institutions)
  Other Names: leuprolide, goserelin, buserelin, or triptorelin
  Arms: Radiation + Androgen Suppression

SUMMARY:
The purpose of this study is to compare the effects, good and/or bad of two treatment methods on subjects and their cancer.

Proton beam radiation therapy is one of the treatments for men with prostate cancer who have localized disease. The benefit of the combination with androgen suppression is not completely understood. This study will compare the use of hypofraction proton therapy (28 treatments) alone to proton therapy with androgen suppression therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate adenocarcinoma (within 365 days of randomization) at intermediate risk for reoccurrence determined by at least one of the following: Gleason Score 7, PSA > = 10 and < = 20, T stage T2b - T2c
* Clinical stages T1-T2c N0 M0 as staged by the treating investigator. (AJCC Criteria 7th Ed.- appendix III).
* Histological evaluation of prostate biopsy with assignment of a Gleason score to the biopsy material; Gleason score must be in the range of 2-7. > 6 cores are strongly recommended.
* PSA values < = 20 ng/ml within 90 days prior to randomization. Obtained prior to biopsy or at least 21 days after prostate biopsy.
* ECOG performance status 0-1 (appendix II) assessed within 90 days of randomization.
* Patients must sign IRB approved study specific informed consent.
* Patients must complete all required pre-entry tests listed in section 4.0 within the specified time frames.
* Patients must be able to start treatment within 56 days of randomization.
* Patients must be at least 18 years old.
* For brachytherapy, an IPSS ≤ 21, or ≤ 17 if patient is on medications to improve urination.
* For brachytherapy, prostate volume must be less than 55cc prior to AS.

Exclusion Criteria:

* Pelvic lymph nodes > 1.5 cm in greatest dimension unless the enlarged lymph node is biopsied and negative.
* Previous prostate cancer surgery to include: prostatectomy, hyperthermia and cryosurgery.
* Previous pelvic radiation for prostate cancer.
* Previous androgen suppression therapy for prostate cancer.
* Active rectal diverticulitis, Crohn's disease affecting the rectum or ulcerative colitis (non-active diverticulitis and Crohn's disease not affecting the rectum are allowed).
* Prior systemic chemotherapy for prostate cancer.
* History of proximal urethral stricture requiring dilatation.
* Current and continuing anticoagulation with warfarin sodium (Coumadin), heparin, low- molecular weight heparin, Clopidogrel bisulfate (Plavix), or equivalent (unless it can be stopped to manage treatment related toxicity or to have a biopsy if needed).
* Major medical, addictive or psychiatric illness which in the investigator's opinion, will prevent the consent process, completion of the treatment and/or interfere with follow-up. (Consent by legal authorized representative is not permitted for this study).
* Evidence of any other cancer within the past 5 years and < 50% probability of a 5 year survival. (Prior or concurrent diagnosis of basal cell or non-invasive squamous cell cancer of the skin is allowed).
* History of myocardial infarction within the last 6 months.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2012-01; Primary Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Morbidity Outcomes | after the initial 100 patients have had a median follow up of at least three years and then every year.
  To determine if androgen suppression along with radiation therapy will result in a higher freedom from failure (FFF) than radiation therapy without androgen suppression.
  Freedom from failure (FFF): The events for FFF will be the first occurrence of clinical failure (local recurrence, regional recurrence, or distant metastasis), biochemical failure by the Phoenix definition (PSA ≥ 2 ng/ml over the current nadir PSA) (45) discounting bounces per investigator discretion, or the start of salvage therapy including androgen suppression

SECONDARY OUTCOMES:
Frequency and severity of grade 2 or higher GU and GI toxicity | At 6 months
  Assessment of grade 2 or higher GU and GI toxicity using CTCAE 4.0 criteria
Frequency and severity of GI and GU toxicity | At 3 years
Incidence of quality of life issues | At completion of radiation therapy
Incidence of Freedom from biochemical failure (FFBF) | At 5 years
Incidence of clinical failure: local and/or distant | At 5 years
Incidence of salvage Androgen Suppression use (SAD) | At 5 years
Incidence of progression free survival: using clinical, biochemical and SAD as events | At 5 years
Incidence of overall survival | At 5 years
Incidence of disease-specific survival | At 5 years
Correlate pathologic and radiologic findings with outcomes | At 5 years
Correlate PSA and free PSA levels with outcomes | At 5 years
Correlate testosterone levels and variation with proton therapy and outcomes | At 5 years
Prospectively collect information that will help to define dose-volume relationships of normal structures with acute and chronic toxicity | At 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Vargas, MD, Principal Investigator — Proton Collaborative Group
Locations (4):
- United States (4):
  - Mayo Clinic, Scottsdale, Arizona
  - Northwestern Medicine Chicago Proton Center, Warrenville, Illinois
  - Oklahoma Proton Center, Oklahoma City, Oklahoma
  - Hampton University Proton Therapy Institute, Hampton, Virginia